CLINICAL TRIAL: NCT02991833
Title: "Developing Of A New Incontinence Care Product, And Investigation Of The Effect Of Its On Perineal Dermatitis in Woman Patients Fecal Incontinence"
Brief Title: Developing Of A New Incontinence Care Product
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Leyla Khorshitd, PROFESSOR DR., Ege University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EGE.0.20.05.00/BOY/1718/99Z
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Incontinence-associated Dermatitis; Nursing Care
Keywords: fecal incontinence; care product; bowel incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Of A New Incontinence Care Product (Experimental): Patients were observed and evaluated daily during the morning care between 08:00 AM - 8:30 AM for a maximum 7 days. The visual scale contrived by (Fader et al.(2003) which is based on International Contact Dermatit Score, was used for graded the severity of IAD. Scoring is is 0-to 4 and when scoring is increased the severity of the IAD increased. To evaluate skin integrity, the perineal skin of the patients was observed every day by researcher and was recorded to the Perineal Skin Integrity Assesment Form. The number of defecation, stool consistency, and the number of care product ( the novel incontinent care product) was observed daily and was recorded to the Patient Observation Form. The main study outcomes was IAD.
  Interventions: Other: A New Incontinence Care Product
- Diaper (Active Comparator): Patients were observed and evaluated daily during the morning care between 08:00 AM - 8:30 AM for a maximum 7 days. The visual scale contrived by (Fader et al.(2003) which is based on International Contact Dermatit Score, was used for graded the severity of IAD. Scoring is is 0-to 4 and when scoring is increased the severity of the IAD increased. To evaluate skin integrity, the perineal skin of the patients was observed every day by researcher and was recorded to the Perineal Skin Integrity Assesment Form. The number of defecation, stool consistency, and the number of care product (diaper ) was observed daily and was recorded to the Patient Observation Form. The main study outcomes was IAD.
  Interventions: Other: Diaper

INTERVENTIONS:
Other: A New Incontinence Care Product — The novel incontinent care product is dressed and removed removed by opening both sides. In the part surrounding the waist and thights of the novel incontinent care product flexibility is achieved by planting rubber bien. When developing new incontinence care products was taken counselling from a faculty member from Department of Textile Engineering of one University Faculty of Engineering. The insurance policies was prepared for each patients attended to the study (Number: 481360).New care product is put on the experimental group. Perineal care was made to patients twice a day and after each defecation. After each perineal care, the novel incontinent care product was changed.
  Arms: Of A New Incontinence Care Product
Other: Diaper — In patients of the diaper group was used the optimum adult diaper (Pads, Linea TENA, SCA, Hygiene, Goteborg, Sweden) which was available in the market. Perineal care was made to patients twice a day and after each defecation. After each perineal care, the diaper was changed.
  Arms: Diaper

SUMMARY:
The aim of this randomized controlled clinical trial, prospective study is to developing a new incontinece care product for containing the fecal incontinence and to examine the effect of this new product on prevention of perineal dermatitis.

DETAILED DESCRIPTION:
Urinary and faecal incontinence which affected the large number of people are common and embarrassing health problems. Urinary incontinence affects the life quality , and causes to isolation and depression. Faecal incontinence can cause to psychosocial problems such as loss of self-esteem, progressive isolation, social stigmatisation and reduces the life quality, also burden a high cost on the patients and the community . Both urinary and fecal incontinence may leads to incontinence-associated dermatitis (IAD), an inflamatory skin disease, which is a a clinical evolution of skin damage associated with moisture , as a result of chronic or repeated exposure of the skin to urine or fecal matter. In IAD shows as redness with or without blistering, erosion, or loss of the skin barrier function IAD which causes discomfort and stres for patients , is a serious and common problem in many health care setting and impacts patients' well-being. Health care professionals who are working in many health institutions struggled to giving the optimal care to keep incontinent patients' skin in a healthy condition. When IAD developed, the risk of infection, the length of hospitalization, and morbidity increases and those patients are at greater risk of developing a pressure ulser.

The research question was; are there differences in the incidence of IAD in patients with fecal incontinence by a new incontinece care versus adult diaper.

ELIGIBILITY:
Inclusion Criteria:

* bedridden patients who had fecal and urinary incontinence,
* had not diabetes mellitus,
* patients whose perineal and perianal skin is intact,
* had indwelling urethral catheter and
* patient who accepted to participate to the study

Exclusion Criteria:

* patients who had diabetes mellitus,
* patients whose had darkly pigmented area in the perineal and perianal area,
* patients had pressure ulcers or erithema
* who have not accepted to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
A New Incontinence Care Product associated dermatitis | 3 months
  Women patients were observed and evaluated daily during the morning care between 08:00 AM - 8:30 AM for a maximum 7 days. The visual scale contrived by (Fader et al.(2003) which is based on International Contact Dermatit Score, was used for graded the severity of IAD. Scoring is is 0-to 4 and when scoring is increased the severity of the IAD increased. To evaluate skin integrity, the perineal skin of the patients was observed every day by researcher and was recorded to the Perineal Skin Integrity Assesment Form. The number of defecation, stool consistency, and the number of care product (diaper and the novel incontinent care product) was observed daily and was recorded to the Patient Observation Form. The main study outcomes was IAD.We defined IAD having an erithema score of 1 or more, in the skin of buttock, sacrum, thight and groin.

SECONDARY OUTCOMES:
Diaper associated dermatitis | 3 months
  Women patients were observed and evaluated daily during the morning care
  between 08:00 AM - 8:30 AM for a maximum 7 days. The visual scale contrived by (Fader et al.(2003) which is based on International Contact Dermatit Score, was used for graded the severity of IAD. Scoring is is 0-to 4 and when scoring is increased the severity of the IAD increased. To evaluate skin integrity, the perineal skin of the patients was observed every day by researcher and was recorded to the Perineal Skin Integrity Assesment Form. The number of defecation, stool consistency, and the number of care product (diaper and the novel incontinent care product) was observed daily and was recorded to the Patient Observation Form. The main study outcomes was IAD.We defined IAD having an erithema score of 1 or more, in the skin of buttock, sacrum, thight and groin.

CONTACTS AND LOCATIONS:
Overall Officials: LEYLA KHORSHID, Professor, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patients were observed and evaluated daily during the morning care between 08:00 AM - 8:30 AM for a maximum 7 daysThe visual scale contrived by (Fader et al.(2003) which is based on International Contact Dermatit Score, was used for graded the severity of IAD. Scoring is is 0-to 4 and when scoring is increased the severity of the IAD increased. Scoring is is 0-to 4 and when scoring is increased the severity of the IAD increased.
Time Frame: 3 months
Access Criteria: perineal dermatitis, fecal incontinence